CLINICAL TRIAL: NCT04620681
Title: CD8 Depleted, Non-Engrafting, HLA Mismatched Unrelated Donor Lymphocyte Infusion in Patients With MDA and Secondary AML
Brief Title: CD8 Depleted, Non-engrafting, HLA Mismatched Unrelated Infusion With MDS and Secondary AML
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MCC-20042; G6095 (Other Grant/Funding Number: FDA)
Record Dates: First submitted 2020-11-03; First posted 2020-11-09 (Actual); Results first posted 2025-10-22 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Myelodysplastic Syndromes; Secondary Acute Myeloid Leukemia
Keywords: MDS; sAML
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1 Dose Level 1 (Experimental): All participants will receive cytotoxic induction chemotherapy with a standard of care cytarabine-based regimen. 24-36 hours after chemotherapy cessation, participants will receive CD8-depleted non-engrafting HLA-mismatched unrelated donor lymphocyte infusion (NE-DLI) at dose level 1: 1X10^6 CD4 T Cells/kg
  Interventions: Biological: CD8 Depleted, Non-engrafting,HLA mismatched unrelated donor lymphocytes; Drug: Standard of Care Chemotherapy
- Phase 1 Dose Level 2 (Experimental): All participants will receive cytotoxic induction chemotherapy with a standard of care cytarabine-based regimen. 24-36 hours after chemotherapy cessation, participants will receive CD8-depleted non-engrafting HLA-mismatched unrelated donor lymphocyte infusion (NE-DLI) at dose level 2: 1X10^7 CD4 T Cells/kg
  Interventions: Biological: CD8 Depleted, Non-engrafting,HLA mismatched unrelated donor lymphocytes; Drug: Standard of Care Chemotherapy
- Phase 1 Dose Level 3 (Experimental): All participants will receive cytotoxic induction chemotherapy with a standard of care cytarabine-based regimen. 24-36 hours after chemotherapy cessation, participants will receive CD8-depleted non-engrafting HLA-mismatched unrelated donor lymphocyte infusion (NE-DLI) at dose level 3: 5 X10^7 CD4 T Cells/kg
  Interventions: Biological: CD8 Depleted, Non-engrafting,HLA mismatched unrelated donor lymphocytes; Drug: Standard of Care Chemotherapy
- Phase 2 -Treatment at Maximum Tolerated Dose (MTD) (Experimental): All participants will receive cytotoxic induction chemotherapy with a standard of care cytarabine-based regimen. 24-36 hours after chemotherapy cessation, participants will receive CD8-depleted non-engrafting HLA-mismatched unrelated donor lymphocyte infusion (NE-DLI) at MTD.
  Interventions: Biological: CD8 Depleted, Non-engrafting,HLA mismatched unrelated donor lymphocytes; Drug: Standard of Care Chemotherapy

INTERVENTIONS:
Biological: CD8 Depleted, Non-engrafting,HLA mismatched unrelated donor lymphocytes — Infusion of mononuclear cells, apheresis products depleted of CD8+ T cells using the CliniMACS® system with CliniMACS® CD8 reagent
Drug: Standard of Care Chemotherapy — Standard of care cytarabine-based chemotherapy

SUMMARY:
The purpose of the study is to determine the safety of an investigational treatment for myelodysplastic syndrome (MDS) after the first therapy (such as azacitidine or decitabine) stops working or after progression of MDS to acute myeloid leukemia (AML). Funding source - FDA OOPD.

DETAILED DESCRIPTION:
The purpose of the study is to determine the safety of an investigational treatment for myelodysplastic syndrome (MDS) after the first therapy (such as azacitidine or decitabine) stops working or after progression of MDS to acute myeloid leukemia (AML).

Patients with advanced MDS are treated with hypomethylating agents (HMAs) such as azacitidine or decitabine. These medications can be effective for a few months to a few years, but usually lose effect eventually. This study is attempting to design a therapy called "non-engrafting, CD8 depleted donor lymphocyte infusion" or "NE-DLI" as a treatment for these diseases.

ELIGIBILITY:
Inclusion Criteria:

Myelodysplastic Syndrome (MDS) having failed hypomethylating agent (HMA) therapy cohort:

* Age 18-79 years, inclusive
* Pathologically confirmed MDS or myelodysplastic/myeloproliferative overlap (MDS/MPN)
* IPSS-R score intermediate, high or very high
* Must have failed therapy with an HMA (defined as lack of response by International Working Group criteria (1) or intolerance of the drug)

Secondary Acute Myeloid Leukemia (sAML):

* Pathologically confirmed AML according to World Health Organization (WHO) criteria
* Evidence of an antecedent hematologic disorder (AHD) prior to acute leukemia including a known prior diagnosis of MDS, MPN or MDS/MPN or data suggestive of an AHD such as cytopenias, fibrosis, macrocytic anemia, cellular or dysplasia at or prior to the time of diagnosis. If available, MDS-defining karyotypes (-7/del(7q), -5/del(5q), del(13q), del(11q), del(12p), t(12p), del(9q), idic(X)(q13), t(17p) (unbalanced translocations) or i(17q) (ie, loss of 17p), t(11;16)(q23;p13.3), t(3;21)(q26.2;q22.1), t(1;3)(p36.3;q21), t(2;11)(p21;q23), inv(3)(q21q26.2), t(6;9)(p23;q34)) or somatic mutations in multiple genes including p53, TET2, JAK2, CALR, MPL, ASXL1, RUNX1, SRSF2, SF3B1, U2AF1, ZRSR2, ASXL1, EZH2, BCOR, or STAG2 would also confirm eligibility.
* Age 60-79 years, inclusive
* May be previously untreated

For both cohorts:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Deemed eligible to receive cytotoxic chemotherapy
* Creatinine clearance (CrCl)>50ml/min
* Total bilirubin <2 mg/dL (except for patients with Gilbert's disease), AST and ALT < 3x ULN
* Left Ventricular Ejection Fraction ≥ 50%
* Willing and able to participate in study assessments

Exclusion Criteria:

* Patients who have had systemic chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier. Hydroxyurea during this period may be given as a bridging therapy to maintain disease stability while awaiting treatment. Intrathecal chemotherapy within this time frame is permitted. Intrathecal chemotherapy may be continued during protocol therapy in order to consolidate or maintain a central nervous system (CNS) remission, but not to treat active CNS disease
* Acute promyelocytic leukemia, or the presence of t(15;17)
* Patients receiving any other investigational agents
* Uncontrolled concurrent illness including, but not limited to, ongoing and uncontrolled infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because there is an unknown but potential risk for adverse events in the fetus. Breastfeeding should be discontinued if the mother is treated. These potential risks may also apply to other agents used in this study
* Patients who have any debilitating medical or psychiatric illness that would preclude their giving informed consent or their receiving optimal treatment and follow-up
* Patients with a poor functional status of ECOG 3-4, or otherwise deemed unfit to tolerate induction chemotherapy.
* Patients with blastic transformation of chronic myelogenous leukemia are ineligible
* Exposure to a humanized mouse chimeric antibody, as this could sensitize patients to components of the CD8 depletion column that may be present in small amounts in the cell product
* Prior allogenic hematopoietic cell transplant

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2024-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Pidala, MD, PhD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Phase 1 Dose Level 1 | Phase 1 Dose Level 2 | Phase 1 Dose Level 3 | Phase 2 -Treatment at Maximum Tolerated Dose (MTD)
Started | 3 | 3 | 3 | 10
Completed | 3 | 3 | 3 | 10
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 Dose Level 1 | Phase 1 Dose Level 2 | Phase 1 Dose Level 3 | Phase 2 -Treatment at Maximum Tolerated Dose (MTD) | Total
Number analyzed (Participants) | 3 | 3 | 3 | 10 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 1 | 4 | 7
  >=65 years | 2 | 2 | 2 | 6 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 1 | 5 | 8
  Male | 1 | 3 | 2 | 5 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 3 | 2 | 2 | 10 | 17
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 3 | 2 | 3 | 10 | 18
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 10 | 19

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of CD8 Depleted Non-engrafting HLA-mismatched Unrelated Donor Lymphocytes Infusion (NE-DLI)
Description: Maximum Tolerated Dose will be determined by testing increasing doses of CD8 depleted non-engrafting HLA-mismatched unrelated donor lymphocytes infusion (NE-DLI).
Time Frame: Up to 60 days per dose level
Measure: Number; unit: 10^7 CD4 cells/kg
Groups:
- Maximum Tolerated Dose (MTD): All participants from dose escalation phase who received treatment at either dose level 1, dose level 2, or dose level 3.
Arm/Group | Maximum Tolerated Dose (MTD)
Number analyzed (Participants) | 9
10^7 CD4 cells/kg | 5

2. Secondary Outcome: Overall Response Rate
Description: Overall Response Rate is defined as Complete Response + Partial Response using RECIST v1.1 criteria.
Time Frame: Up to 12 months
Population: As specified in the protocol, only participants treated at the MTD are included in this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of Participants with Response
Groups:
- Participants Treated at MTD: Participants treated at MTD.
Arm/Group | Participants Treated at MTD
Number analyzed (Participants) | 13
percentage of Participants with Response | 61.5 [31.6 to 86.1]

3. Secondary Outcome: Progression Free Survival
Description: Progression Free Survival is defined as the time from enrollment to date of progression or death, or censor at last follow-up date.
Time Frame: Up to 12 months
Population: As specified in the protocol, only participants treated at the MTD are included in this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Participants Treated at MTD
Number analyzed (Participants) | 13
Months | 8.7 [1.4 to NA] — Not reached

4. Secondary Outcome: Overall Survival
Description: Overall Survival is defined as the time from study enrollment to death from any cause or censored at last follow up date
Time Frame: Up to 12 months
Population: As specified in the protocol, only participants treated at the MTD are included in this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Participants Treated at MTD
Number analyzed (Participants) | 13
Months | 11.9 [2.5 to NA] — Not Reached

5. Secondary Outcome: Hematologic Response
Description: Hematologic response will be determined using International Working Group 2006 criteria for MDS patients and the International Working Group 2003 criteria for AML
Time Frame: Up to 12 months
Population: As specified in the protocol, only participants treated at the MTD are included in this outcome measure.
Measure: Number; unit: Number of Participants achieving CR
Groups:
- Participants Treated at MTD - sAML: Participants Treated at MTD - sAML
- Participants Treated at MTD - MDS: Participants Treated at MTD - MDS
Arm/Group | Participants Treated at MTD - sAML | Participants Treated at MTD - MDS
Number analyzed (Participants) | 11 | 2
Number of Participants achieving CR | 7 | 0

ADVERSE EVENTS:
Time Frame: 1 Year
Arm/Group | Phase 1 Dose Level 1 | Phase 1 Dose Level 2 | Phase 1 Dose Level 3 | Phase 2 -Treatment at Maximum Tolerated Dose (MTD)
All-Cause Mortality (participants affected / at risk) | 3/3 | 3/3 | 2/3 | 5/10
Serious Adverse Events (participants affected / at risk) | 2/3 | 0/3 | 3/3 | 1/10
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Dose Level 1 (N=3) | Phase 1 Dose Level 2 (N=3) | Phase 1 Dose Level 3 (N=3) | Phase 2 -Treatment at Maximum Tolerated Dose (MTD) (N=10)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Dose Level 1 (N=3) | Phase 1 Dose Level 2 (N=3) | Phase 1 Dose Level 3 (N=3) | Phase 2 -Treatment at Maximum Tolerated Dose (MTD) (N=10)
Anemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (5) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endocarditis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 3 (3) | 2 (2) | 4 (5)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Platelet count decreased (Investigations) | 2 (4) | 1 (3) | 1 (2) | 2 (9)
White blood cell decreased (Investigations) | 3 (4) | 0 (0) | 0 (0) | 1 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (6) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-29): https://cdn.clinicaltrials.gov/large-docs/81/NCT04620681/Prot_SAP_000.pdf